CLINICAL TRIAL: NCT01669291
Title: Effect of GnRH Antagonist Protocol vs Agonist Long Protocol During Controlled Hyperstimulation (COH)for Assisted Reproduction on IVF Outcome, Peak Estradiol Level, and Duration of Stimulation.
Brief Title: Effect of GnRH Antagonist vs Agonist Long on IVF Outcome, Peak Estradiol Level,and Duration of Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Main Line Fertility Center (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MLFC-003
Record Dates: First submitted 2012-08-09; First posted 2012-08-21 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Fertility
MeSH Terms: interventions — Urofollitropin; Menotropins; Leuprolide; ganirelix; cetrorelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bravelle & Menopur Agonist Long Protocol (Active Comparator): Patients will use an LH agonist (Lupron) starting on day 18 of the oral contraceptive pill (OCP), 5 units b.i.d. followed by 5 units q.d. beginning on day one of stimulation medications. The 5 units q.d. dose will continue until the day of hCG administration.Patients will administer Bravelle and Menopur for ovarian stimulation.
  Interventions: Drug: Bravelle and Menopur; Drug: Agonist
- Bravelle & Menopur Antagonist Protocol (Active Comparator): Patients will complete standard dose of oral contraceptive pill (OCP) and will then administer GnRH antagonist (ganirelix acetate or cetrorelix acetate) 0.25 mg q.d. during the stimulation phase when the lead follicle size reaches 12mm. The antagonist will continue until the day of hCG administration. Patients will administer Bravelle and Menopur for ovarian stimulation.
  Interventions: Drug: Bravelle and Menopur; Drug: Antagonist

INTERVENTIONS:
Drug: Bravelle and Menopur — Bravelle and Menopur are used for controlled ovarian stimulation (COH)
Drug: Agonist — Agonist (Lupron) is used to suppress endogenous pituitary LH for the premature LH surges.
  Other Names: Leuprolide Acetate; Lupron
  Arms: Bravelle & Menopur Agonist Long Protocol
Drug: Antagonist — Ganirelix acetate or cetrorelix acetate Agonist is used to suppress endogenous pituitary LH for the premature LH surges.
  Other Names: ganirelix acetate; cetrorelix acetate
  Arms: Bravelle & Menopur Antagonist Protocol

SUMMARY:
The purpose of this study is to determine if utilizing GnRH antagonists versus agonist long protocol during controlled ovarian stimulation (COH) with human-derived gonadotropins for assisted reproduction affects IVF outcome, peak estradiol level, and duration of stimulation.

DETAILED DESCRIPTION:
No detailed description

ELIGIBILITY:
Inclusion Criteria:

* Ages 21-40 (inclusive up to 41)
* Day 2-4 FSH < or equal to 10
* Antimullerian Hormone (AMH) greater than or equal to 1.0
* Between 5 and 20 antral follicles on day 2-4
* Body Mass Index (BMI)>or equal to 18 and < or equal to 32

Exclusion Criteria:

* Smokers
* Polycystic Ovarian Disease
* Endometriosis greater than Stage I
* Testicular aspirated sperm

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2012-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
To determine if COH in IVF patients using Bravelle & Menopur with antagonists results in improved or equal IVF results compared to patients using agonist. | One year

SECONDARY OUTCOMES:
To determined if COH in IVF patients using Bravelle & Menopur with antagonists results in lower peak estradiol levels compared to agonist | One year
To determine if COH patients using Bravelle & Menopur with antagonist antagonists results inn shorter period of stimulation compared with agonist. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Glassner, M.D., Principal Investigator — Main Line Fertility Center; Sharon H. Anderson, Ph.D, Study Director — Main Line Fertility Center
Locations (1):
- Main Line Fertility Center, Bryn Mawr, Pennsylvania, United States

REFERENCES:
- [Background] Ludwig, Michael. GnRH antagonists. Textbook of Assisted Reproductive Technologies - Laboratory and Clinical Perspectives. Third edition. Edited by Gardner, D, Weissman, A, Howles, C, Shoham, Z. 2009: 539-552.
- [Background] Ludwig M, Katalinic A, Diedrich K. Use of GnRH antagonists in ovarian stimulation for assisted reproductive technologies compared to the long protocol. Meta-analysis. Arch Gynecol Obstet. 2001 Nov;265(4):175-82. doi: 10.1007/s00404-001-0267-2. PMID 11789740
- [Background] Fluker M, Grifo J, Leader A, Levy M, Meldrum D, Muasher SJ, Rinehart J, Rosenwaks Z, Scott RT Jr, Schoolcraft W, Shapiro DB; North American Ganirelix Study Group. Efficacy and safety of ganirelix acetate versus leuprolide acetate in women undergoing controlled ovarian hyperstimulation. Fertil Steril. 2001 Jan;75(1):38-45. doi: 10.1016/s0015-0282(00)01638-1. PMID 11163814
- [Background] Ludwig M, Felberbaum RE, Devroey P, Albano C, Riethmuller-Winzen H, Schuler A, Engel W, Diedrich K. Significant reduction of the incidence of ovarian hyperstimulation syndrome (OHSS) by using the LHRH antagonist Cetrorelix (Cetrotide) in controlled ovarian stimulation for assisted reproduction. Arch Gynecol Obstet. 2000 Jul;264(1):29-32. doi: 10.1007/pl00007479. PMID 10985616